CLINICAL TRIAL: NCT02269683
Title: Randomized Controlled Trial of Robotic vs. Laparoscopic Distal Pancreatectomy for Pancreatic Cancer - The DAVID-study
Brief Title: Robotic vs. Laparoscopic Distal Pancreatectomy for Pancreatic Cancer
Acronym: DAVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTG-02
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot-assisted (Experimental): Distal pancreatectomy via robot-assisted minimally-invasive approach
  Interventions: Procedure: Robot-assisted distal pancreatectomy
- Laparoscopic (Active Comparator): Distal pancreatectomy via a conventional laparoscopic approach
  Interventions: Procedure: Laparoscopic distal pancreatectomy

INTERVENTIONS:
Procedure: Robot-assisted distal pancreatectomy
  Arms: Robot-assisted
Procedure: Laparoscopic distal pancreatectomy
  Arms: Laparoscopic

SUMMARY:
The present randomized controlled trial evaluates the incidence of R1 resections in patients undergoing robotic distal pancreatectomy compared to the laparoscopic technique.

DETAILED DESCRIPTION:
Surgical resection the only potentially curative therapeutic approach in patients with pancreatic cancer. Among the clinicopathologic factors that are associated with long-term survival, a complete (i.e. R0) tumor resection is of utmost significance. Numerous reports have already demonstrated detection of tumor cells at the resection margin on microscopic examination (i.e. R1 resection) is associated with poor long-term survival. However, studies using a standardized pathological work-up of operative specimen from patients with pancreatic cancer revealed that most pancreatic resections are R1 resections. Innovative surgical techniques that reduce the incidence of R1 resections may provide a promising approach to improve the outcome of patients with pancreatic cancer.

For patients requiring a distal pancreatectomy, a laparoscopic pancreatic resection is increasingly performed, as it may enhance postoperative recovery without compromising oncological safety compared to the open approach. However, laparoscopic technique does not affect the proportion of patients with complete (R0) resections. Furthermore, the inability to control major vasculature frequently results in conversion to the open approach. The vast majority of R1 margins are located at the retroperitoneal dissection surface. Due to technical limitations, the open and the laparoscopic technique may not further reduce the incidence of positive resection margins at this location.

The 3D visualization provided by the robotic approach together with improved dexterity of the surgeon are likely to enable a meticulous dissection at the posterior dissection margin. This may result in a significant reduction of patients with positive resection margins. However, to date there has been no randomized controlled trial that compared the robotic to the laparoscopic technique. As health-care interventions need to prove efficacy and safety in well-designed randomized controlled trials, the present randomized controlled trial was designed to test, if robotic distal pancreatectomy increases the incidence of patients with complete (R0) tumor resection for pancreatic cancer. Secondary endpoints include oncological parameters such as the number of harvested lymph nodes and factors of perioperative outcome such as perioperative complications (Clavien-Dindo classification), pancreatic fistula, in-hospital mortality, blood loss and conversion rates.

ELIGIBILITY:
Inclusion Criteria:

* Suspected malignant disease of the pancreas scheduled for distal pancreatectomy
* Patient eligible for laparoscopic resection
* ≥ 18 years of age
* Written informed consent

Exclusion Criteria:

* Planned multi-visceral and/or vascular resection
* Evidence of distant metastases
* Expected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
R1 resection rate | 10 days
  Proportion of patients with complete macroscopic resection, but microscopic residual tumour. Pathological evaluation will be performed by experienced, board-certified pathologists using standardized protocols according to current guidelines. Importantly, pathologists will be blinded for patients treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, University Hospital Dresden, Dresden, Germany